CLINICAL TRIAL: NCT02327039
Title: The Effects of Dapagliflozin on HDL Particles Subtypes and Reverse Cholesterol Transport in Type 2 Diabetic Patients. A 12 Weeks Randomized Placebo-controlled Phase IV Study
Brief Title: The Effects of Dapagliflozin on HDL Particles Subtypes and Reverse Cholesterol Transport in Type 2 Diabetic Patients
Acronym: DAPA-HDL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Azienda Ospedaliera di Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3302/AO/14; 2014-004270-42 (EudraCT Number); ESR-14-10088 (Other Grant/Funding Number: Astrazeneca)
Record Dates: First submitted 2014-12-15; First posted 2014-12-30 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10 mg tablet once daily for 12 weeks
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo 10 mg tablet once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Sodium glucose cotransporter-2 inhibitor
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Placebo — Tables of Dapagliflozin placebo
  Arms: Placebo

SUMMARY:
In Phase 2b/3 clinical trials, Dapagliflozin has been shown to raise HDL cholesterol levels by about 4 mg/dl (1 mmol/l), which is generally considered a clinically-meaningful change. As this HDL cholesterol increase is carried out with concomitant improvement in glucotoxicity and body weight reduction, it is possible that treatment with Dapagliflozin also improves HDL function. This is important because clinical, epidemiological and experimental studies indicate that HDL function may be more important than HDL cholesterol levels in determining the protective cardiovascular effects of HDL particles. In addition, knowing the effects of Dapagliflozin on HDL function can help interpreting the increase in HDL cholesterol levels observed in Dapagliflozin-treated patients. Finally, discovery of extra-glycemic effects of Dapagliflozin will shed new light on the potential benefits of therapy with Dapagliflozin and SGLT2i in general. So far, no study evaluated the effects of Dapagliflozin (or other SGLT2i) on HDL function.

The investigators hypothesize that Dapagliflozin, in addition to raising HDL cholesterol levels, also increases HDL functionality, measured as reverse cholesterol transport and anti-oxidant capacity, in patients with T2DM

DETAILED DESCRIPTION:
Sodium glucose co-transport-2 (SGLT-2) inhibitors (SGLT-2i), a new class of glucose-lowering agents, reduce tubular glucose reabsorption, thus lowering blood glucose without stimulating insulin release. SGLT-2i have been found to be effective in improving glucose control in type 2 diabetic patients at any disease stage, and also when added to insulin in type 1 diabetic patients. In addition to the glycosuric effect, SGLT-2i reduce body weight and blood pressure and determine an increase in HDL cholesterol levels. HDL mediate reverse cholesterol transport, by extracting cholesterol from peripheral tissues and cells and vehiculating it to the liver. This function, which is regulated that by enzyme cholesteryl esther transfer protein (CETP), is considered a fundamental mechanism of protection from accumulation of cholesterol in the vasculature and a physiologic barrier against atherosclerosis development and protection. The sophisticated method to precisely assess reverse cholesterol transport in vitro are available in our research lab. Although it has been reported that therapy with SGLT-2i raise HDL concentrations by about 4 mg/dL (0.1 mmol/L), the mechanisms remains unclear and it is important to assess whether or not this quantitative increase is coupled to functional improvement in reverse cholesterol transport. In fact, previous studies on HDL-raising therapies have clarified that not all HDL particles and functional and HDL cholesterol levels might not be representative of the reverse cholesterol transport processes. In addition to cholesterol transport, normal HDL particles also have anti-oxidant and anti-inflammatory properties, that are important to translate HDL cholesterol levels into cardiovascular protection. Several HDL subclasses have been identified, having different composition and anti-atherosclerotic properties.

Dapagliflozin (Bristol-Myers Squibb Company [BMS]-512148) is a highly potent, selective, and reversible inhibitor of sodium-glucose cotransporter 2 (SGLT2), the major transporter responsible for renal glucose reabsorption. Dapagliflozin lowers plasma glucose by inhibiting the renal reabsorption of glucose and by promoting its urinary excretion. A tablet formulation of dapagliflozin for oral administration has been approved in over 40 countries including the European Union (EU) and the United States (US) and is under review in numerous countries around the world. Dapagliflozin is approved by AIFA with determination number 909/2013 dated 16/10/2013, and marketing authorization number 042494070/E. In the Phase 2b and 3 program, dapagliflozin has been studied as monotherapy and in combination with metformin, pioglitazone, glimepiride, sitagliptin, and insulin. As of 15-Nov-2012 (date of most recent pooled analysis), a total of 9,412 subjects with T2DM were treated in 16 Phase 3, double-blind, controlled clinical studies conducted to evaluate the safety and efficacy of dapagliflozin; 5,952 subjects in these studies were treated with dapagliflozin for up to 80 weeks. The Phase 2b and 3 program established that dapagliflozin is effective in reducing HbA1c in a broad range of subjects regardless of disease progression/duration or concomitant use of antidiabetic therapies. Improvements in glycemic control were seen when dapagliflozin was given as monotherapy; as add-on combination therapy to sitagliptin or metformin, to sulfonylurea (glimepiride), to thiazolidinedione (pioglitazone), or to insulin (± oral antidiabetic drugs [OADs]); or as initial combination therapy with metformin.

HDL levels and function. Observational studies provide overwhelming evidence that a low high-density lipoprotein (HDL)-cholesterol level increases the risk of coronary events, both in healthy subjects and in patients with coronary heart disease. Based on in vitro experiments, several mechanistic explanations for the atheroprotective function of HDL have been suggested. The HDL functions currently most widely held to account for the antiatherogenic effect include participation in reverse cholesterol transport, protection against endothelial dysfunction, and inhibition of oxidative stress. Yet, several recent pharmacological and genetic studies have failed to demonstrate that increased plasma levels of HDL-C resulted in decreased cardiovascular disease risk, giving rise to a controversy regarding whether plasma levels of HDL-C reflect HDL function, or that HDL is even as protective as assumed. The evidence from preclinical and clinical studies shows that HDL can promote the regression of atherosclerosis when the levels of functional particles are increased from endogenous or exogenous sources. The data show that regression results from a combination of reduced plaque lipid and macrophage contents, as well as from a reduction in its inflammatory state. Although more research will be needed regarding basic mechanisms and to establish that these changes translate clinically to reduced cardiovascular disease events, that HDL can regress plaques suggests that the recent trial failures do not eliminate HDL from consideration as an atheroprotective agent but rather emphasizes the important distinction between HDL function and plasma levels of HDL-C. While HDL from healthy subjects can directly stimulate endothelial cell production of nitric oxide and anti-inflammatory, anti-apoptotic, and anti-thrombotic effects as well as endothelial repair processes, growing evidence suggests that the vascular effects of HDL can be highly heterogeneous and vasoprotective properties of HDL are altered in patients with coronary disease. In fact, HDL has been shown to undergo a loss of function in several pathophysiological states, as in the acute phase response, obesity and chronic inflammatory diseases. Some of these diseases were also shown to be associated with increased risk for cardiovascular disease. One such disease that is associated with HDL dysfunction and accelerated atherosclerosis is diabetes mellitus, a disease in which the HDL particle undergoes diverse structural modifications that result in significant changes in its function, such as glycation and oxidation.

In Phase 2b/3 clinical trials, Dapagliflozin has been shown to raise HDL cholesterol levels by about 4 mg/dl (1 mmol/l), which is generally considered a clinically-meaningful change. As this HDL cholesterol increase is carried out with concomitant improvement in glucotoxicity and body weight reduction, it is possible that treatment with Dapagliflozin also improves HDL function. This is important because clinical, epidemiological and experimental studies indicate that HDL function may be more important than HDL cholesterol levels in determining the protective cardiovascular effects of HDL particles. In addition, knowing the effects of Dapagliflozin on HDL function can help interpreting the increase in HDL cholesterol levels observed in Dapagliflozin-treated patients. Finally, discovery of extra-glycemic effects of Dapagliflozin will shed new light on the potential benefits of therapy with Dapagliflozin and SGLT2i in general. So far, no study evaluated the effects of Dapagliflozin (or other SGLT2i) on HDL function.We hypothesize that Dapagliflozin, in addition to raising HDL cholesterol levels, also increases HDL functionality, measured as reverse cholesterol transport and anti-oxidant capacity, in patients with T2DM.

This will be a randomized, placebo controlled, parallel group study in 36 type 2 diabetic patients to assess the effects of Dapagliflozin on HDL levels and function.

The general objective of the project is to detect a significant differences in the changes versus baseline of the patients' HDL cholesterol efflux capacity, HDL levels, HDL subclasses, HDL anti-oxidant activity, CETP activity, serum/plasma cytokines and adipokines (IL-6, IL-8, PAI-1, TNF-α, visfatin, resistin, adiponectin, leptin) in patients randomized to dapagliflozin compared to those randomized to placebo

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Female and male subjects aged 18-75 years
* Type 2 diabetes on oral agents +/- insulin
* Diabetes duration >6 months
* HbA1c 7.0-10.0%

Exclusion Criteria:

* Acute illness or infection
* Recent (within 1 month) surgery, trauma, cardiovascular event
* Recent (within 3 months) variation of statin therapy/dose
* Therapy with HDL-modifying drugs, such as fibrates, omega-3 fatty acids, and niacin
* Alcoholism
* Very high baseline HDL levels (>90 mg/dL)
* Previous history of recurrent (≥2 episodes) urinary tract infections or genital infections (a single remote episode not to be considered an exclusion criterion)
* History of hypotension, episodes of volume depletion / dehydration.
* Chronic renal failure (eGFR<60 ml/min/1.73 mq)
* Chronic liver disease (SGOT or GPT >2-fold ULN, or cirrhosis)
* Elevated hematocrit (>50% for men or >45% for women)
* Heart failure, NYHA classes III-IV
* Hypersensitivity to Dapagliflozin or its excipients
* Treatment with pioglitazone or GLP-1 receptor agonists
* Women with childbearing potential

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in reverse cholesterol transport, measured as cholesterol efflux capacity of patient's plasma | 12 weeks
  Detection of a significant change in reverse cholesterol transport by patients' plasma in Dapagliflozin compared to placebo-treated diabetic patients.
  The cholesterol efflux capacity of patient's plasma will be measured as arbitrary units using radioactive cholesterol loaded macrophages

SECONDARY OUTCOMES:
Changes from baseline in HDL cholesterol levels | 12 weeks
  Detection of significant changes in Dapagliflozin compared to placebo-treated T2D patients in HDL cholesterol levels, measured by standard chemistry in patients' serum
Changes from baseline in the distribution in HDL subclasses | 12 weeks
  Detection of significant changes in Dapagliflozin compared to placebo-treated T2D patients in the distribution of HDL subclasses (% distribution in each of the 10 HDL subclasses, measured with the Lipoprint system)
Changes from baseline in HDL antioxidant activity | 12 weeks
  Detection of significant changes in Dapagliflozin compared to placebo-treated T2D patients in the HDL antioxidant activity, measured as serum concentrations of paraoxonase 1 (PON1), PON1 activity and TBARS.
Changes from baseline in CETP activity | 12 weeks
  Detection of significant changes in Dapagliflozin compared to placebo-treated T2D patients in CETP activity, determined as U/ml using a commercially available assay
Safety as measured by monitoring of adverse events | 12 weeks
  Safety and tolerability will be assessed during the study according to the protocol for monitoring of adverse events. Number of adverse events will be collected for each group

OTHER OUTCOMES:
Exploratory analyses - changes from baseline in plasma cytokines | 12 weeks
  Detection of significant changes in Dapagliflozin compared to placebo-treated T2D patients of the plasma concentrations of the following factors: IL-6, IL-8, PAI-1, TNF-α, visfatin, resistin, adiponectin, leptin, measured using multiplex arrays.
Exploratory analyses - changes from baseline in plasma bioimpedance body composition | 12 weeks
  Detection of significant changes in Dapagliflozin compared to placebo-treated T2D patients of fat mass, fat-free mass and water, as determined by bioimpedance analysis.
Exploratory analyses - changes from baseline in impedance cardiography analysis | 12 weeks
  Detection of significant changes in Dapagliflozin compared to placebo-treated T2D patients of heart rate; stroke volume; cardiac output; acceleration index; velocity index; systolic time ratio; left ventricular ejection time; left cardiac work; left cardiac work index; systemic vascular resistance; thoracic fluid content; total arterial compliance

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Metabolic Diseases, University Hospital of Padova, Padua, Italy

REFERENCES:
- [Derived] Bonora BM, Vigili de Kreutzenberg S, Avogaro A, Fadini GP. Effects of the SGLT2 inhibitor dapagliflozin on cardiac function evaluated by impedance cardiography in patients with type 2 diabetes. Secondary analysis of a randomized placebo-controlled trial. Cardiovasc Diabetol. 2019 Aug 14;18(1):106. doi: 10.1186/s12933-019-0910-5. PMID 31412874
- [Derived] Fadini GP, Bonora BM, Zatti G, Vitturi N, Iori E, Marescotti MC, Albiero M, Avogaro A. Effects of the SGLT2 inhibitor dapagliflozin on HDL cholesterol, particle size, and cholesterol efflux capacity in patients with type 2 diabetes: a randomized placebo-controlled trial. Cardiovasc Diabetol. 2017 Apr 4;16(1):42. doi: 10.1186/s12933-017-0529-3. PMID 28376855